CLINICAL TRIAL: NCT06567145
Title: Assessing the Effectiveness and Feasibility of Group-based Treatment for Self-stigma in People With Mental Disorders: a Pragmatic Multisite Randomized Controlled Trial in Routine Mental Health Services in North-east Italy
Brief Title: A Group-based Treatment for Self-stigma in People With Mental Disorders in North-east Italy
Acronym: NECT-ITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Antonio Lasalvia, Associate Professor of Psychiatry at the Department of Neurosciences, Biomedicine, and Movement Sciences, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 358CET
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Stigma; Mental Disorders; Self-stigma
Keywords: stigma; narrative enhancement cognitive therapy; narrative therapy; cognitive therapy; mental disorders; self-stigma
MeSH Terms: conditions — Social Stigma; Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrative Enhancement and Cognitive Therapy (NECT) (Experimental): Patients assigned to the experimental gropu will receive the Narrative Enhancement and Cognitive Therapy (NECT), a structured psychological intervention aimed at reducing self-stigma in individuals with severe mental illness. It was developed in early 2000s in the USA by Philip Yanos, David Roe and Paul Lysaker. Patients in the experimental group will also receive routine treatment typically provided within their usual care settings.
  Interventions: Behavioral: Narrative Enhancement Cognitive Therapy (NECT)
- Control group (No Intervention): Patients in the control group will continue to receive the routine treatment typically provided within their usual care settings, which usually includes pharmacological treatment + outpatient visits (for monitoring pharmacological treatment and symptom management) + (if needed) other psychosocial treatments (e.g., individual or group therapy, family psychoeducation, cognitive rehabilitation, job placements/supported employment).

INTERVENTIONS:
Behavioral: Narrative Enhancement Cognitive Therapy (NECT) — The Narrative Enhancement and Cognitive Therapy (NECT) consists of 20 group sessions divided into five parts: orientation (2 sessions), psychoeducation on stigma (3 sessions), cognitive restructuring (7 sessions), narrative enhancement (7 sessions), and a concluding reflection (1 session). The program helps participants challenge self-stigmatizing beliefs, develop coping skills, and create a new, positive narrative about themselves. Each session lasts about an hour, with a structured format of introduction, main discussion, and conclusion, encouraging active participation and reflection on personal experiences. The intervention ultimately fosters self-efficacy, control, and hope for the future.
  Arms: Narrative Enhancement and Cognitive Therapy (NECT)

SUMMARY:
Self-stigma refers to the internalization of negative stereotypes by individuals with mental disorders, leading to beliefs that they are dangerous, aggressive, or incapable of working. This phenomenon has harmful effects on various aspects of life, such as adherence to treatment, self-esteem, quality of life, and can increase feelings of despair and suicide risk. To address these issues, the Narrative Enhancement and Cognitive Therapy (NECT) was developed. NECT is a group-based intervention consisting of 20 sessions designed to reduce self-stigma in individuals with mental disorders.

This study aims to evaluate the efficacy and feasibility of NECT in 416 patients from 26 mental health centers in Northeast Italy. It is structured as a pragmatic, multicenter, randomized controlled trial with two parallel arms. The study will assess the impact of NECT on several psychological dimensions, including levels of self-stigma, self-esteem, hope, empowerment, perception of recovery, mental well-being, and stigma-related stress. The findings of this research are expected to contribute to the understanding of effective treatments for patients with mental disorders, particularly those burdened by high levels of self-stigma, and to improve their recovery outcomes.

DETAILED DESCRIPTION:
BACKGROUND Population surveys indicate that people generally hold distorted views and negative stereotypes about individuals suffering from mental disorders. For example, 60% of the population believes that patients with mental disorders are aggressive or violent, and 50% believe they are incapable of working. Research has also found that most individuals with mental disorders are aware of the presence of these stereotypes in society, and over 70% expect to be treated unjustly by others because of their condition. Additionally, 60-70% of patients with mental disorders believe that most people would refuse to have someone with a mental disorder as a friend, neighbor, colleague, or partner. While some individuals with mental disorders may react to these stereotypes with indifference or anger, most end up accepting these stereotypes as true, internalizing them and attributing them to themselves; this phenomenon is known as internalized stigma or self-stigma. One of the largest studies in this field estimated that 41% of individuals with schizophrenia spectrum disorders experience high levels of self-stigma. Other studies have reported similar rates. The literature has found that self-stigma is associated with worse recovery outcomes. A recent meta-analysis reports significant correlations between self-stigma and a lack of hope, self-esteem, and self-efficacy, poorer subjective quality of life, greater symptom severity, and lower treatment adherence. Self-stigma can be both a consequence and a cause of negative outcomes. When self-stigma plays a causal role, it can become a target for treatment. Yanos and colleagues proposed the illness identity model which provides a set of detailed and testable hypotheses regarding the potential causal role that self-stigma plays in influencing recovery outcomes in individuals with mental disorders. This model suggests that when identity is influenced by self-stigma, individuals believe that recovery is not possible, reducing hope (i.e., expectations about one future) and self-esteem. Despair and low self-esteem, in turn, increase the risk of suicide, reduce social interaction, lead to the use of passive coping strategies for symptoms, and reduce treatment adherence. As patients use avoidant coping strategies, they may also lose their jobs. Finally, avoidant coping, social isolation, and reduced social functioning can increase the severity of psychotic symptoms. Empirical support for this model comes from the findings of two studies conducted by different research groups. Building on the evidence of the role that self-stigma plays in recovery processes, Narrative Enhancement and Cognitive Therapy (NECT) was developed as a treatment protocol aimed at reducing self-stigma in individuals with mental disorders. NECT is a structured group treatment that combines psychoeducation (to help participants challenge stigmatizing beliefs about mental illness and recovery with empirical and scientific data), cognitive restructuring (aimed at teaching skills to modify negative beliefs about oneself related to stigma), and narrative enhancement (designed to help participants improve their ability to integrate themes like trust and self-worth into their narratives). To date, five studies have tested the effectiveness of NECT. The first, conducted in the United States with a small group of 39 patients, failed to highlight significant effects of NECT on self-stigma, likely due to the small sample size; however, the intervention was found to be feasible and well-tolerated by participants. A study conducted in Israel with 119 patients showed that participation in the NECT program was associated with significant improvements in self-esteem, quality of life, and hope. Similarly, a randomized controlled trial with a 6-month follow-up conducted in Gothenburg, Sweden, found that the NECT intervention was associated with significant improvements in self-esteem and self-stigma, and that these improvements were maintained at six months. A subsequent randomized controlled study conducted in the United States with 170 patients with schizophrenia spectrum disorders demonstrated that NECT could produce significant improvements in self-stigma and other variables, including avoidant coping, compared to the supportive control intervention. Finally, a randomized controlled trial implemented in Taiwan showed more significant results from NECT in improving self-esteem and reducing perceived discrimination compared to the control intervention. These studies demonstrate that NECT's effectiveness is supported by robust empirical evidence, qualifying it as an evidence-based intervention and suggesting its large-scale implementation. Unfortunately, in Italy, interventions against self-stigma in individuals with mental disorders are not regularly provided. Where anti-self-stigma interventions are offered, they are generally not based on solid evidence of effectiveness. This delay is due to the unavailability of manualized interventions, such as NECT, in our language. Moreover, the anti-self-stigma interventions published in the literature have so far been tested in geographical contexts and within healthcare organizations very different from those in our country. Therefore, it is unclear how these interventions, if made available in Italian, could be applicable within our healthcare settings.

OBJECTIVES The objectives of this study are: (1) to evaluate the effectiveness of this approach in the clinical routine of mental health centers; (2) to test the feasibility of the new Italian version of the NECT treatment in patients who seek care at mental health centers in a large area of north-eastern Italy. Overall, this project will enhance knowledge of optimal treatments for patients with mental disorders burdened by high self-stigma, with the aim of improving their recovery outcomes. The study is a pragmatic, multicenter, randomized controlled trial with two parallel arms: intervention group and control group.

INTERVENTIONS The intervention group will receive Narrative Enhancement and Cognitive Therapy (NECT), a structured group therapy aimed at reducing self-stigma in individuals with severe mental disorders. NECT, originally developed by Philip Yanos and colleagues, has been adapted into Italian for this study and consists of 20 sessions divided into five parts: orientation, psychoeducation, cognitive restructuring, narrative enhancement, and conclusion. Each part is designed to help participants reflect on their experiences, challenge self-stigmatizing beliefs, and foster a new, positive identity. The control group will continue with their usual care, which typically involves a combination of pharmacological treatment and psychosocial interventions provided by public mental health services. The study will systematically collect information about the care received by participants during the trial.

STUDY DURATION AND RANDOMIZATION PROCEDURE NECT sessions during approximately one hour, structured into an introduction, a central discussion, and a conclusion. The NECT intervention is considered an add-on treatment, meaning participants will continue receiving their standard care in addition to the group therapy. The control group will continue with their usual treatment, which may include medication, symptom management, and psychiatric rehabilitation. Staff involved in delivering the NECT intervention will undergo specific training to ensure consistent and effective implementation.

Treatment fidelity will be monitored through audio recordings of selected sessions, evaluated using the NECT Fidelity Scale.

The study also includes a feasibility assessment, measuring participant engagement, session completion rates, and feedback from both participants and facilitators to identify factors that may impact the implementation of NECT in clinical settings.

The study is designed to be completed over 12 months. It begins with protocol approval, followed by a two-month recruitment phase to enroll eligible participants. Once recruitment is complete, a five-month intervention phase will take place, during which participants will undergo the NECT treatment. The final five months are allocated for data entry, analysis, and the preparation of results for publication.

The study involves 26 community mental health centers (CMHCs) across the Veneto region, the Trento province, and the city of Bolzano.

The randomization process is crucial for ensuring the validity of the trial. Each CMHC will recruit 16 patients, for a total of 416 participants. They will be randomly assigned to either the NECT intervention group or a control group, maintaining a 1:1 allocation ratio.

This stratified randomization by CMHC ensures that the unique characteristics of each center are accounted for, contributing to the robustness of the study's findings. The randomization will be carried out using specialized software to ensure fairness and consistency across all centers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years or older.
2. Individuals must have a diagnosis of schizophrenia, schizoaffective disorder, schizoid disorder, schizophreniform disorder, bipolar I or II disorder, or major depressive disorder, according to DSM-5 criteria.
3. Participants must be outpatients with clinical stability for at least 3 months, with no changes in pharmacological treatment during this period.
4. Participants must have sufficient knowledge of written and spoken Italian.
5. Participants must score above 1 on the ISMI (Internalized Stigma of Mental Illness) scale, indicating at least moderate levels of self-stigma.

Exclusion Criteria:

1. Individuals unable to provide informed consent are excluded.
2. Participants with intellectual disabilities are excluded.
3. Individuals with primary diagnosis of personality disorder or substance dependence condition are excluded.
4. Participants engaged in other programs that could influence self-stigma (e.g., social cognitive rehabilitation, social skills training) during the study are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Differences in the level of self-stigma | From enrollment to the end of treatment at 20 weeks
  The primary outcome of the study is the differences in the level of self-stigma (or internalized stigma) between the group receiving the NECT (Narrative Enhancement and Cognitive Therapy) intervention and the control group. These differences will be assessed using the total score from the ISMI (Internalized Stigma of Mental Illness) scale. The ISMI (Internalized Stigma of Mental Illness) scale is a 29-item self-report questionnaire used to measure self-stigma in individuals with mental illness. It includes five subscales: Alienation, Stereotype Endorsement, Discrimination Experience, Social Withdrawal, and Stigma Resistance. Higher scores indicate greater internalized stigma. The measurements will be taken at two time points: at baseline (T0) and at the end of the treatment (T1). The main objective is to observe the change in the total ISMI score over time, comparing the two groups to evaluate the effectiveness of the NECT intervention in reducing self-stigma.

SECONDARY OUTCOMES:
Self-esteem | From enrollment to the end of treatment at 20 weeks
  The Rosenberg Self Esteem Scale (RSES) is used to assess self-esteem, a key indicator of a person's overall sense of self-worth. The scale consists of 10 items rated on a 4-point Likert scale, ranging from "strongly agree" to "strongly disagree." Higher scores reflect greater self-esteem. This outcome aims to evaluate whether the NECT intervention improves participants' self-perception and confidence from baseline (T0) to the end of the treatment (T1). Self-esteem is crucial for mental health, influencing motivation, resilience, and overall well-being, making it a vital measure of the intervention's effectiveness.
Hope and expectations about the future | From enrollment to the end of treatment at 20 weeks
  Hope is measured using the Beck Hopelessness Scale (BHS-9), which assesses an individual's negative expectations about the future. This 9-item self-report questionnaire asks participants to respond to statements with "true" or "false," providing a total score that indicates the level of hopelessness. Higher scores signify greater hopelessness. This outcome seeks to determine whether the NECT intervention can increase participants' sense of hope and optimism about their future, a critical factor in recovery from mental illness. Enhanced hope can lead to better coping strategies, increased motivation, and improved overall mental health.
Empowerment | From enrollment to the end of treatment at 20 weeks
  Empowerment is measured through the Boston University Empowerment Scale (BUES), which captures the degree to which individuals feel in control of their lives and capable of influencing their own recovery. The BUES is a 28-item self-report scale with items rated on a 4-point Likert scale. It includes five subscales: anger, optimism and control over the future, self-esteem/self-efficacy, power/perceived loss of power, and community activism and autonomy. Higher scores indicate greater empowerment. This outcome evaluates whether NECT enhances participants' feelings of empowerment, which is crucial for taking an active role in their recovery and improving their quality of life.
Recovery Perception | From enrollment to the end of treatment at 20 weeks
  The Recovery Assessment Scale (RAS) is used to measure participants' perceptions of their own recovery. This scale includes 20 items distributed across five factors: personal confidence and hope, willingness to ask for help, goal orientation and success, reliance on others, and not being dominated by symptoms. Participants rate their agreement with these statements on a 5-point Likert scale. Higher scores indicate a stronger sense of recovery. This outcome assesses whether the NECT intervention helps participants perceive themselves as more recovered, which is essential for their long-term mental health and well-being.
Mental wellbeing | From enrollment to the end of treatment at 20 weeks
  Mental well-being is assessed using the Warwick and Edinburgh Mental Wellbeing Scale (WEMWBS), which measures positive mental health through 14 items. These items are rated on a 5-point Likert scale, with higher scores indicating better mental well-being. The scale captures aspects such as positive thoughts, feelings, and psychological functioning. This outcome aims to determine if the NECT intervention can enhance participants' overall mental well-being, including their ability to function effectively in daily life and experience positive emotions, which are vital components of recovery from mental illness.
Stigma as a stressor | From enrollment to the end of treatment at 20 weeks
  The Stigma Stress Scale is used to evaluate the extent to which stigma is perceived as a stressor by the participants. This scale comprises two items: one measuring the perceived harm due to stigma and the other assessing the resources available to cope with it. Responses are given on a 7-point Likert scale, and the difference between the two scores represents the level of stigma-related stress. Higher scores indicate greater stress. This outcome seeks to assess whether the NECT intervention can reduce the stress associated with stigma, which is crucial for improving mental health and reducing the burden of self-stigma on daily life.
Screening rate | From enrollment to the end of treatment at 20 weeks
  The number of patients who meet the ISMI screening criteria compared to those who meet the inclusion and exclusion criteria.
Eligible rate | From enrollment to the end of treatment at 20 weeks
  The number of eligible patients who agree to participate in the study.
Intervention completion rate | From enrollment to the end of treatment at 20 weeks
  The number of participants who completed the intervention, the reasons for participant dropout.
Exposure rate | From enrollment to the end of treatment at 20 weeks
  The proportion of participants "exposed" to the intervention, defined as attending at least six sessions or completing one of the key phases: psychoeducation, cognitive restructuring, or narrative enhancement.
Perceptions of Implementation Factors | From enrollment to the end of treatment at 20 weeks
  In this outcome, open-ended questions will be utilized to gather detailed insights from participants and facilitators. These questions are designed to encourage respondents to express their thoughts, experiences, and opinions freely, providing a deeper understanding of the factors that may facilitate or hinder the implementation of the intervention. By using open-ended questions, the aim is to capture a wide range of perspectives and nuanced feedback that might not be fully addressed through closed-ended questions alone.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata (AOUI) Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymzed cumulative indivudual participant data (IPD) will be made available upon reasonable request by writing an e-mail to the PI (Prof. Antonio Lasalvia)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available after the publication of the main paper
Access Criteria: Write an e-mail to antonio.lasalvia@univr.it

REFERENCES:
- [Background] Huang LT, Liu CY, Yang CY. Narrative enhancement and cognitive therapy for perceived stigma of chronic schizophrenia: A multicenter randomized controlled trial study. Arch Psychiatr Nurs. 2023 Jun;44:59-68. doi: 10.1016/j.apnu.2023.04.004. Epub 2023 Apr 15. PMID 37197864
- [Background] Yanos PT, Lysaker PH, Silverstein SM, Vayshenker B, Gonzales L, West ML, Roe D. A randomized-controlled trial of treatment for self-stigma among persons diagnosed with schizophrenia-spectrum disorders. Soc Psychiatry Psychiatr Epidemiol. 2019 Nov;54(11):1363-1378. doi: 10.1007/s00127-019-01702-0. Epub 2019 Apr 1. PMID 30937510
- [Background] Hansson L, Lexen A, Holmen J. The effectiveness of narrative enhancement and cognitive therapy: a randomized controlled study of a self-stigma intervention. Soc Psychiatry Psychiatr Epidemiol. 2017 Nov;52(11):1415-1423. doi: 10.1007/s00127-017-1385-x. Epub 2017 Apr 19. PMID 28424854
- [Background] Cavelti M, Rusch N, Vauth R. Is living with psychosis demoralizing? Insight, self-stigma, and clinical outcome among people with schizophrenia across 1 year. J Nerv Ment Dis. 2014 Jul;202(7):521-9. doi: 10.1097/NMD.0000000000000160. PMID 24933416
- [Background] Yanos PT, Roe D, Lysaker PH. The Impact of Illness Identity on Recovery from Severe Mental Illness. Am J Psychiatr Rehabil. 2010 Apr;13(2):73-93. doi: 10.1080/15487761003756860. PMID 20802840
- [Background] Livingston JD, Boyd JE. Correlates and consequences of internalized stigma for people living with mental illness: a systematic review and meta-analysis. Soc Sci Med. 2010 Dec;71(12):2150-61. doi: 10.1016/j.socscimed.2010.09.030. Epub 2010 Oct 12. PMID 21051128
- [Background] Brohan E, Elgie R, Sartorius N, Thornicroft G; GAMIAN-Europe Study Group. Self-stigma, empowerment and perceived discrimination among people with schizophrenia in 14 European countries: the GAMIAN-Europe study. Schizophr Res. 2010 Sep;122(1-3):232-8. doi: 10.1016/j.schres.2010.02.1065. Epub 2010 Mar 26. PMID 20347271
- [Background] Lasalvia A, Zoppei S, Van Bortel T, Bonetto C, Cristofalo D, Wahlbeck K, Bacle SV, Van Audenhove C, van Weeghel J, Reneses B, Germanavicius A, Economou M, Lanfredi M, Ando S, Sartorius N, Lopez-Ibor JJ, Thornicroft G; ASPEN/INDIGO Study Group. Global pattern of experienced and anticipated discrimination reported by people with major depressive disorder: a cross-sectional survey. Lancet. 2013 Jan 5;381(9860):55-62. doi: 10.1016/S0140-6736(12)61379-8. Epub 2012 Oct 18. PMID 23083627
- [Background] Pescosolido BA, Medina TR, Martin JK, Long JS. The "backbone" of stigma: identifying the global core of public prejudice associated with mental illness. Am J Public Health. 2013 May;103(5):853-60. doi: 10.2105/AJPH.2012.301147. Epub 2013 Mar 14. PMID 23488508
- [Background] Angermeyer MC, Dietrich S. Public beliefs about and attitudes towards people with mental illness: a review of population studies. Acta Psychiatr Scand. 2006 Mar;113(3):163-79. doi: 10.1111/j.1600-0447.2005.00699.x. PMID 16466402
- [Derived] Lasalvia A, Bodini L, Cristofalo D, Fin V, Yanos PT, Bonetto C. Assessing the effectiveness and the feasibility of a group-based treatment for self-stigma in people with mental disorders in routine mental health services in North-East Italy: study protocol for a pragmatic multisite randomized controlled trial. Trials. 2025 Jan 31;26(1):35. doi: 10.1186/s13063-025-08739-4. PMID 39891254